

**CorEvitas Statistical Analysis Plan (SAP):** Treatment Patterns and 6-Month Effectiveness of Tofacitinib in CorEvitas' Rheumatoid Arthritis Registry



**NOTE**: Final SAP revised to include descriptive data on history of biologics presented by MOA and clarification regarding study population for looking at outcomes.

# 1. Table of Contents

| Section | | Page |
|------------|--------------------------------------|--------------|
| 1. Table o | of Contents | 2 |
| 2. Resear | rch Protocol | 3 |
| 2.1. Bac | ckground and Rationale | 3 |
| 2.2. Obj | jectives | 3 |
| 2.2.1. | Objective 1 | 3 |
| 2.2.2. | Objective 2 | 3 |
| 2.2.3. | Objective 3 | 3 |
| 2.3. Hyp | pothesis | 3 |
| 2.4. Res | search Design | 3 |
| 2.4.1. | Study Type | 3 |
| 2.4.2. | Data Source | 3 |
| 2.4.3. | Study Populations | 2 |
| 2.4.4. | Sample Size and Power Considerations | 2 |
| 2.4.5. | Time Periods | 5 |
| 2.4.6. | Variables | <del>6</del> |
| 2.5. Plai | n of Analysis | 8 |
| 2.5.1. | Descriptive analysis | 9 |
| 2.5.2. | Effectiveness Analysis | 9 |
| 3. Shell T | ables | 11 |

## 2. Research Protocol

## 2.1. Background and Rationale

Previous work in the Corrona registry described the early experience of tofacitinib (tofa) initiators. As tofa has been on the market since 2012, it is possible that there has been a shift to use of tofa as an earlier line of therapy. Therefore, there is a need to update the analyses of treatment patterns and effectiveness. This query will inform the design of future comparative effectiveness analyses.

## 2.2. Objectives

To describe treatment patterns and effectiveness of tofa initiators in the Corrona RA registry.

## 2.2.1. Objective 1

To describe the demographics, clinical characteristics, and treatment patterns of tofa initiators at time of initiation.

## 2.2.2. Objective 2

To estimate 6-month effectiveness in tofa initiators.

## 2.2.3. Objective 3

To estimate 12-month effectiveness in tofa initiators.

## 2.3. Hypothesis

This is a descriptive query, thus there are no a priori hypotheses.

## 2.4. Research Design

## 2.4.1. Study Type

This study is a retrospective observational study using registry data for RA patients.

## 2.4.2. Data Source

Corrona<sup>1</sup> was founded in 2000 and is an independent registry without any ownership links to the pharmaceutical industry. This registry contains clinical data (e.g. disease activity scores, laboratory results, comorbidities, imaging results, patient-reported outcomes data, etc.) that is not available in claims databases such as the Truven MarketScan database. The Corrona RA

registry is the largest longitudinal registry studying chronic diseases in the world. The current Corrona dataset includes 189 private and academic active clinical sites with over 800 physicians throughout 42 states in the U.S. The Corrona Rheumatoid Arthritis study is an ongoing longitudinal clinical registry that was established in 2001. This registry collects data from both the physicians and the patients at the time of a regular office visit. Corrona has enrolled over 54,000 patients with RA. The collection of data from Corrona represents over 195,000 patient years of data.

To be enrolled in the registry, patients must meet the following criteria:

- Have RA diagnosed by a rheumatologist
- Be at least 18 years of age
- Must be able and willing to provide informed consent

## 2.4.3. Study Populations

#### Inclusion Criteria

For this analysis patients must:

- 1. Initiate tofa (defined as first ever use of tofa) at the Corrona enrollment visit or at a Corrona follow up visit from November 2012 onward.
- 2. Have CDAI measured at baseline.
- 3. Have a 6-month or 12-month follow-up visit and CDAI measured at 6-month or 12-month follow-up visit

Note: Additionally, the specified populations will be used to calculate each of the following variables.

- Achievement of LDA (CDAI≤10).
  - Among patients with moderate or high disease activity (CDAI>10) at baseline.
- Rate of response at follow up visit-achievement of remission (CDAI≤2.8).
  - Among patients with LDA, moderate, or high disease activity (CDAI>2.8) at baseline.
- Achievement of LDA or remission defined by DAS28(ESR) (<= 3.2)</li>
  - o Among patients who have DAS28>3.2 at the initiation visit.
- Achievement of "mild pain", defined as ≤ 20mm on 100 VAS scale
  - o Among patients who have pain >20 mm on 100 VAS at the initiation visit

## **2.4.4.** Sample Size and Power Considerations

#### Sample size

As of the end of August 31, 2020, there are 2744 RA patients who initiated tofa in the Corrona RA registry. Of these, 1650 have a visit at 6 months (3-9 months) and 1223 have a visit at 12

months (10-15 months) have CDAI measured at the initiation visit (baseline) and at 6- or 12-month follow-up visit.

Number of initiators with tofa initiation and had a 6-month or 12-month follow up visit in 4 milestones

| | With 6 month<br>Follow up | With 12 month<br>Follow up |
|--------------|---------------------------|----------------------------|
| Milestone 1 | | |
| Monotherapy | 730 | 536 |
| Combotherapy | 920 | 687 |
| Total | 1650 | 1223 |
| Milestone 2 | | |
| 2nd line | 236 | 168 |
| 3rd line | 333 | 234 |
| 4+ line | 1027 | 781 |
| Total | 1596 | 1183 |
| Milestone 3 | | |
| 5 mg/ BID | 732 | 579 |
| 11 mg/QD | 663 | 463 |
| Total | 1395 | 1042 |
| Milestone 4 | | |
| 2012-2014 | 451 | 349 |
| 2015-2017 | 725 | 597 |
| 2018-2020 | 474 | 277 |
| Total | 1650 | 1223 |

### **Definition of line of therapy:**

1<sup>st</sup> line: no prior use of any DMARD at time of initiation

2<sup>nd</sup> line: prior use of at least one csDMARD and no prior use of any biologic

3<sup>rd</sup> line: prior use of at least one csDMARD and prior use of 1 biologic

4<sup>th</sup> line+: prior use of at last one csDMARD and prior use of 2+ biologics

### 2.4.5. Time Periods

## Study visits

The Corrona RA registry is an observational registry collecting patient and physician data at regular patient clinical visits with the rheumatologist. Unlike in clinical trials, visits are not timed at exact uniform time periods. We will define the 6-month visit as a Corrona visit that occurs between 3-9 months post- index visit. We will define the 12 month visit as a Corrona visit that occurs between 10-15 months post index visit. If the patient had more than one visit in the

window between 3 and 9 months (or 10-15 months), the visit closest to 6 (or 12) months will be selected.

## 2.4.6. Variables

### For Objective 1 (Demographics, clinical characteristics, treatment patterns):

Demographic/socioeconomic characteristics

Age, sex, race, education, work status, insurance

#### Lifestyle

Weight, body mass index(BMI), smoking status

### History of comorbidities

- History of CV disease (include the following: MI, stroke, acute coronary syndrome, coronary artery disease, CHF, revascularization procedure including percutaneous coronary intervention [PCI], coronary artery bypass grafting [CABG] or coronary artery stents, ventricular arrhythmia, cardiac arrest, unstable angina, peripheral ischemia, peripheral arterial disease, hypertension, other CV, DVT, and TIA.)
- History of malignancy (breast cancer, lung cancer, lymphoma, skin cancer, other cancer)
- History of hypertension, diabetes, osteoporosis, fibromyalgia, and depression

#### Clinical Characteristics and Assessments

- Duration of disease
- Age of onset
- CDAI (continuous, categorical)
- Tender joint count (28)
- Swollen Joint count (28)
- Physician global assessment (0-100)
- DAS28(ESR)
- Patient global assessment (0-100)
- Patient reported pain (0-100)
- Patient reported fatigue (0-100)
- HAQ (0-3)
- mHAQ
- Morning stiffness (yes/no)
- Morning stiffness duration (hours)

### Treatment Characteristics and Medication history

 Concomitant therapies (Monotherapy, Combo with: MTX alone, other CDMARD, MTX + other CDMARD)

- Number of prior biologics/JAKis (TNFi: Enbrel, Humira, Remicade, Cimzia, Simponi; non-TNFi: Orencia, Actemra, Rituxan, Kineret, Kevzara; JAKis: Olumiant, Rinvoq)
- Number of prior csDMARDs (MTX, Arava, Azulfidine, Plaquenil, Cyclosporine, Imuran, Minocin, Cuprimine, Ridaura)
- Steroid use
  - History of prednisone use (yes/no)
  - Current prednisone use (yes/no)
  - Prednisone dose (in users)
- Mode of Action (MOA) History
  - TNF inhibitor
  - Non-TNF inhibitor
  - csDMARDs
  - o tsDMARDs
- History of treatment of MOA (Ever)
  - TNF inhibitor
  - Non-TNF inhibitor
  - o csDMARDs
  - o tsDMARDs

### Reason for initiation of Tofa:

- Number of patients with at least 1 initiation reason reported
- Total number of reasons
- o % Safety, % Efficacy, % Cost/Insurance, %Other reasons

#### Reason for Discontinuation of tofa (Among those who discontinue at or before 6-months):

- o Total number (%) of discontinuations
- o Number of patients with at least 1 reason reported
- Total number of reasons
- % Safety, % Efficacy, % Cost/Insurance, %Other reasons

### For objective 2 (6-months effectiveness) and objective 3 (12-months effectiveness)

### Primary outcomes:

• Achievement of LDA (CDAI ≤ 10)

#### Secondary outcomes:

- Achievement of remission (CDAI ≤ 2.8)
- Δ CDAI
- Δ HAQ

- Δ patient pain
- Δ patient fatigue
- Achievement of mACR20/50/70
- Achievement of LDA or remission defined by DAS28(ESR) (<= 3.2)</li>
- Achievement of "mild pain", defined as ≤ 20mm on 100 VAS scale

## 2.5. Plan of Analysis

### **Definitions:**

<u>Index visit (Baseline)</u>: The Corrona visit with the first reported use of tofa.

Disease activity measures and patient-reported outcomes (PROs) from the index (baseline) visit will be used if the initiation date is the same as the visit date. If tofa is initiated between visits, and the prior visit is within 4 months of the initiation date, disease activity measures and PROs from the prior visit will be used as the baseline value.

## Line of therapy:

1st line: no prior use of any DMARD at time of initiation
2nd line: prior use of at least one csDMARD and no prior use of any biologic
3rd line: prior use of at least one csDMARD and prior use of 1 biologic
4th line+: prior use of at last one csDMARD and prior use of 2+ biologics

## Study Cohorts:

- Overall tofa initiators who meet inclusion criteria
- Tofa monotherapy at initiation visit (tofa only)
- Tofa combo therapy at initiation visit (tofa+MTX, Arava, Azulfidine, Plaquenil, or cyclosporine)
- Tofa initiators by line of therapy in 2<sup>nd</sup> line, 3<sup>rd</sup> line and 4<sup>th</sup> line
- Tofa dose of 5mg, twice a day at initiation visit
- Tofa dose of 11mg, once a day at initiation visit
- Tofa initiators by year of initiation (2012-2014, 2015-2017, 2018-2020)

#### This project will be separated into 4 milestones:

- 1. Analysis in overall tofa initiators, and monotherapy v. combination therapy
- 2. Analysis by line of therapy in 2<sup>nd</sup> line, 3<sup>rd</sup> line and 4<sup>th</sup> line
- Analysis by tofa dose (5mg v. 11mg)
- 4. Analysis by three time periods of initiation (2012-2014, 2015-2017, 2018-2020)

## 2.5.1. Descriptive analysis

Baseline patient demographics and clinical characteristics of (listed in section 2.4.4) will be presented. For categorical variables, n(%) will be presented, and for continuous variables, means, standard deviation (SD), median, 25<sup>th</sup> and 75ths quartile values will be presented in overall tofa initiators, and by group (for each milestone). P-values will be estimated using student-t test for continuous variables between two comparison groups, one-way Anova for continuous variables among three comparison groups and chi-square test for categorical variables. Two sets of baseline tables will be reported – one for patients with 6 months follow-up and one for patients with 12 months follow-up.

## 2.5.2. Effectiveness Analysis

## Primary outcome analyses

We will estimate the rate of response at 6 and 12 months. Response is defined as the achievement of LDA (CDAI≤10) in patients with moderate or high disease activity (CDAI>10) at baseline. Patients who discontinue tofa within 6 (or 12) months and switch to another biologic or JAK will be considered "non-responders". Effectiveness outcomes at the 6- and 12- month visits will be estimated in overall tofa initiators and by groups for each milestone. We will report the rate of response and 95% CI for the proportion of response, for patients overall and for each group in table 5.

### Secondary outcomes analysis

The following secondary outcomes will be considered:

- Rate of response at follow up visit-achievement of remission (CDAI≤2.8) in patients with LDA, moderate, or high disease activity (CDAI>2.8) at baseline. Patients who discontinue tofa within 6 months and switch to another biologic or JAK will be considered "nonresponders".
- Mean of change in CDAI from baseline to follow up visit (6/12). Change in CDAI will be calculated by subtracting baseline CDAI from CDAI measured at 6 months. If a patient discontinues tofa but does not switch to another biologic, the CDAI value at follow up visit (6/12) will be used. If a patient discontinues tofa and switches to another biologic or JAK, the CDAI value at the switch visit will be used for change in CDAI calculation.
- HAQ (HAQ):
   Mean change of HAQ from index date to follow-up visit

- Patient pain (0-100 VAS scale):
   Mean change in pain from index date to follow-up visit
- Patient fatigue (0-100 VAS scale):
   Mean change in fatigue from index date to follow-up visit
- Achievement of modified ACR (mACR)20, mACR50, mACR70
- Achievement of LDA or remission defined by DAS28(ESR) (<= 3.2) in those patients who have DAS28>3.2 at the initiation visit
- Achievement of "mild pain", defined as ≤ 20mm on 100 VAS scale in those patients who have pain >20 mm on 100 VAS at the initiation visit

Mean changes, rates of response, and corresponding 95% confidence intervals will be reported in total and in each group [Table 5].

Two sets of analyses will be report based on patient with 6 month follow up and patients with 12 months follow up.

All statistical analyses will be performed using STATA Version 15.1 (StataCorp, LLC, College Station, TX).

## 3. Shell Tables

Milestone 1: Results for tofa monotherapy and combination therapy

Milestone 2: Results for line of therapy (2<sup>nd</sup>, 3<sup>rd</sup>, 4<sup>th</sup> line)

Milestone 3: Results for tofa dose (5mg and 11mg)

Milestone 4: Results for tofa initiation time periods (2012-2014, 2015-2017, and 2018-2020)

Table 1. Demographic and clinical characteristics at tofa initiation visit, overall and for monotherapy and combination therapy in patients with 6 months follow up.

| | All Patients | Tofa<br>monotherapy | Tofa<br>combination<br>therapy <sup>‡</sup> | <i>P</i> -value* |
|---|---|---|---|---|
| | N= | N= | N= | |
| Demographic/socioeconomic | | | | |
| characteristics | | | | |
| Age: Mean±SD | | | | |
| Median (IQR) | | | | |
| Female: n(%) | | | | |
| Race/Ethnicity: n(%) | | | | |
| White | | | | |
| Hispanic | | | | |
| Black | | | | |
| Asian | | | | |
| Other | | | | |
| Type of Insurance: | | | | |
| None: n (%) | | | | |
| Private: n (%) | | | | |
| Medicare: n (%) | | | | |
| Medicaid: n (%) | | | | |
| Final education: n(%) | | | | |
| Primary | | | | |
| High school | | | | |
| College/Univ. | | | | |
| Unknown | | | | |
| Work Status: n(%) | | | | |
| Full Time | | | | |
| Part Time | | | | |
| Disabled | | | | |

<sup>\*</sup> T-tests will be used to evaluate mean differences between groups for continuous variables, and Chi-square tests will be used to evaluate differences between treatment groups for categorical variables

<sup>\*\*</sup> included: MI, stroke, TIA acute coronary syndrome, coronary artery disease, CHF, revascularization procedure including percutaneous coronary intervention [PCI], coronary artery bypass grafting [CABG] or coronary artery stents, ventricular arrhythmia, cardiac arrest, unstable angina, other CVs, carotid artery disease.

<sup>\*\*\*</sup> History of lung cancer, breast cancer, lymphoma, skin cancer (melanoma and squamous), and other cancer

<sup>‡</sup> Combination therapy refers to tofa+MTX, arava, azulfidine, plaquenil, or cyclosporine

Table 2. RA disease characteristics, disease activity measures and PROs at tofa initiation visit, overall and for monotherapy and combination therapy in patients with 6 months follow up.

| | All Patients | Tofa<br>Monotherapy | Tofa<br>Combination | P value* |
|---|---|---|---|---|
| | | | Therapy <sup>‡</sup> | |
| B4 # | N= | N= | N= | |
| RA disease characteristics | | | | |
| Duration of RA: Mean±SD | | | | |
| Median (IQR) | | | | |
| Age onset RA: Mean±SD | | | | |
| Median (IQR) | | | | |
| Disease Activities | | | | |
| CDAI: Mean±SD | | | | |
| Median (IQR) | | | | |
| Category of disease activity: n(%) | | | | |
| Remission | | | | |
| LDA | | | | |
| MDA | | | | |
| HAD | | | | |
| Tender Joint Count (28): Mean±SD | | | | |
| Median (IQR) | | | | |
| Swollen Joint Count (28): Mean±SD | | | | |
| Median (IQR) | | | | |
| Physician Global Assessment(0-100): | | | | |
| Mean±SD | | | | |
| Median (IQR) | | | | |
| DAS28(ESR): Mean±SD | | | | |
| Median (IQR) | | | | |
| Patient reported outcomes | | | | |
| Patient Global Assessment: Mean±SD | | | | |
| Median (IQR) | | | | |
| Patient Pain Assessment: Mean±SD | | | | |
| Median (IQR) | | | | |
| Patient Fatigue Assessment: Mean±SD | | | | |
| Median (IQR) | | | | |
| HAQ (0-3): Mean±SD | | | | |
| Median (IQR) | | | | |
| mHAQ: Mean±SD | | | | |
| Median (IQR) | | | | |
| Morning Stiffness: n(%) | | | | |

| Stiffness(mins): Mean±SD** |
|------------------------------------|
| Median (IQR) |
| Treatment |
| Concomitant therapies: n(%) |
| None |
| MTX only |
| nonMTX csDMARD only |
| MTX & nonMTX csDMARD |
| History of csDMARD: n(%) |
| None |
| 1 |
| 2+ |
| History of biologics: n(%) |
| None |
| 1 |
| 2+ |
| Prednisone |
| History of prednisone use: n(%) |
| Current prednisone use: n(%) |
| Dose in users: Mean±SD |
| Median (IQR) |
| Mode of Action (MOA) History |
| Immediately previous treatment |
| TNF inhibitor |
| Non-TNF inhibitor |
| csDMARDs |
| tsDMARDs |
| History of treatment of MOA (Ever) |
| TNF inhibitor |
| Non-TNF inhibitor |
| csDMARDs |
| tsDMARDs |

<sup>\*</sup> T-tests will be used to evaluate mean differences between groups for continuous variables, and Chi-square tests will be used to evaluate differences between categorical variables

<sup>\*\*</sup> in patients reported morning stiffness

<sup>‡</sup> Combination therapy refers to tofa+MTX, arava, azulfidine, plaquenil, or cyclosporine

Table 3. Reasons for initiation of tofacitinib in patients with 6 month follow up

| n(%) | All Tofa | Tofa mono | Tofa combo |
|---|---|---|---|
| (,,, | N= | N= | N= |
| # of initiations | | | |
| # of patients reporting at least one reason | | | |
| Total # of reasons | | | |
| Safety | | | |
| Efficacy | | | |
| Cost/Insurance | | | |
| Other reason | | | |

Table 4. Reasons for discontinuation of tofacitinib in 6 months

| n(%) | All | Tofa mono | Tofa combo |
|---------------------------------------------|-----|-----------|------------|
| (70) | N= | N= | N= |
| # of discontinuations | | | |
| # of patients reporting at least one reason | | | |
| Total # of reasons | | | |
| Safety | | | |
| Efficacy | | | |
| Cost/Insurance | | | |
| Other reason | | | |

#### Notes:

- Side effect: includes infection, lymphoma/malignancy, toxicity, serious and minor side effect;
- Efficacy: includes lack of efficacy, disease flare, active disease, primary loss of efficacy, and secondary loss of efficacy, inadequate initial response, failure to maintain initial response;
- Cost/Insurance: includes lack of insurance
- Other reason: includes no longer needed, formulary restriction, patient preference, recent journal report, recent meeting report, withdrawn by FDA, physician preference, peer suggestion, fear of future side effect, patient doing well, and frequency of administration, temporary interruption, to improve compliance, to improve tolerability, route of administration.

Table 5. Outcome measures at 6 months after tofa initiation, overall and for monotherapy and combination therapy groups

| Binary outcomes | All Tofa Initiators | Tofa Monotherapy | Tofa Combo therapy |
|---|---|---|---|
| n(%) | N= | N= | N= |
| 95% CI | | IN- | |
| | n= | n= | n= |
| LDA (CDAI≤10)ª | | | |
| | n= | n= | n= |
| Remission (CDAI≤2.8)b | | | |
| mACR20 | | | |
| mACR50 | | | |
| mACR70 | | | |
| | n= | n= | n= |
| DAS28(ESR)≤3.2 <sup>c</sup> | | | |
| | n= | n= | n= |
| Achievement of "mild pain"<br>(≤ 20mm on 100 VAS) <sup>d</sup> | | | |
| Continue outcomes: | | | |
| Mean (SD) | | | |
| 95% CI | | | |
| Δ CDAI: | | | |
| Δ patient global | | | |
| Δ HAQ | | | |
| Δ patient pain | | | |
| Δ patient fatigue | | | |

<sup>&</sup>lt;sup>a</sup> Calculated among those patients with moderate or high disease activity (CDAI>10) at baseline.

<sup>&</sup>lt;sup>b</sup> Calculated among those patients with LDA, moderate or high disease activity (CDAI>2.8) at baseline.

<sup>&</sup>lt;sup>c</sup> Calculated among those patients who have DAS28>3.2 at the initiation visit

<sup>&</sup>lt;sup>d</sup> Calculated among those patients who have pain >20 mm on 100 VAS at the initiation visit

Tables 6-10 will repeat tables 1-5, by line of therapy (2<sup>nd</sup> line, 3<sup>rd</sup> line, and 4<sup>th</sup> line) for Milestone 2.

Table 11-15 will repeat table 1-5, by tofa dose (5mg/bid and 11mg/qd) for Milestone 3.

Table 16-20 will repeat table 1-5 for the three time periods of initiation (2012-2014, 2015-2017, 2018-2020) for milestone 4.

Table 21-40 will repeat tables 1-20 for patients with 12 months follow up by 4 milestone.

# **Document Approval Record**

**Document Name:** A3921379 Non Interventional Statistical Analysis Plan\_1 April 2020\_re

vised 23 April 2021

**Document Title:** A3921379 Non Interventional Statistical Analysis Plan\_1 April 2020\_re

vised 23 April 2021

Signed By: Date(GMT) Signing Capacity

PPD 17-Aug-2021 04:52:06 Business Line Approver